CLINICAL TRIAL: NCT04378699
Title: Comparison of 2 Neurofeedback Protocols in the Treatment of Attention Deficit Hyperactivity Disorder in Children and Adolescents
Brief Title: 2 Neurofeedback Protocols in the Treatment of Attention Deficit Hyperactivity Disorder in Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-HPNCL-03
Record Dates: First submitted 2017-11-07; First posted 2020-05-07 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: ADHD
Keywords: ADHD; neurofeedback
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: single-center interventional biomedical research with direct individual benefit, randomized with two active arms (without placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMR Sensory Motor Rhythm (12-15 Hz) (Experimental): 3 X 10 SMR workout sessions (12-15 Hz) C4 unipolar placement, central region
  Interventions: Other: SMR (12-15 Hz)
- the alpha band (8 -12Hz) (Experimental): 3 x 10 training sessions of the higher frequencies of the alpha band (8 -12Hz), unipolar placement Fz, fronto-central region
  Interventions: Other: alpha band (8 -12Hz)

INTERVENTIONS:
Other: SMR (12-15 Hz) — SMR training sessions (12-15 Hz) C4 unipolar placement, central region
  Arms: SMR Sensory Motor Rhythm (12-15 Hz)
Other: alpha band (8 -12Hz) — 3 x 10 training sessions of the higher frequencies of the alpha band (8 -12Hz), unipolar placement Fz, fronto-central region
  Arms: the alpha band (8 -12Hz)

SUMMARY:
Attention Deficit Disorder with or without Hyperactivity (ADD / H) is a public health problem since it has short and long-term consequences, affects about 5% of children of school age but remains unknown and therefore under- diagnostic.

The investigator will performed a controlled and randomized research to compare the effects of two neurofeedback protocols on the repercussions of Attention Deficit AD / Hyperactivity Disorder (HD) symptoms, in particular the hyperactivity on which the improvements reported in the literature are less with usual protocols.

DETAILED DESCRIPTION:
Attention deficit disorder with or without hyperactivity (ADD / H) is a public health problem since it has short and long-term consequences, affects about 5% of children of school age but remains unknown and therefore under- diagnostic. In the symptomatic triad of inattention, impulsivity and hyperactivity, there is often a psychopathological disorder, a learning and / or sleep disorder. Medication treatment with methylphenidate is the reference in terms of prescription to reduce the symptoms of AD / HD. However, the limitations of its long-term effectiveness, tolerance of side effects, and parental distrust of psychostimulant treatment are gradually opening the door to new therapeutic approaches.

Neurofeedback is considered by the scientific world as a promising and effective neurocognitive learning technique in the treatment of Attention Deficit Disorder with Hyperactivity ADHD and several neurological and psychiatric disorders. Its principle is to increase the patient's ability to regulate his own brain activity, captured by an ElectroEncephaloGram (EEG), after visual and auditory feedback.

In this controlled and randomized research, the investigator will compare the effects of two neurofeedback protocols on the repercussions of AD / HD symptoms, in particular the hyperactivity on which the improvements reported in the literature are less with usual protocols.

Seventy children and adolescents aged 7 to 15 in two groups will benefit from thirty neurofeedback sessions each, either on a so-called Sensory Motor Rhythm (SMR) protocol or on a protocol called Upper Alpha. To date, no studies have identified the effects of a NF Upper Alpha protocol on improving sleep, hyperactivity and comorbidities in patients with ADHD in a controlled and randomized manner. nor on personality dimensions related to the processes of self-regulation of the patient involved in Neurofeedback (NF) treatment.

The investigator expects superior clinical improvement of ADHD symptoms and sleep disorders in the NF upper alpha training group in patients not following any parallel drug or therapy regimen. The investigator expects stability of the effects of treatment after several months of stopping neurofeedback sessions, without taking or recovery of psychostimulant.

This research protocol would make it possible for dozens of children and adolescents to benefit from an alternative treatment (in the absence of placebo conditions) in order to achieve a clinical improvement of at least 30% of their patients. symptoms related to AD / HD, as well as to develop a field of research still little investigated in France. On the other hand, parents would be more likely to accept effective neurofeedback treatment than psychostimulant treatment, especially since it may have side effects. In addition, the validation of clinical improvements following a neurofeedback protocol aimed at increasing the relative power of alpha waves at frontal sites would be encouraging for clinical practice and future research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Children or teenagers between 8 and 15 years old included
* Subject with mixed-type ADHD (attention deficit hyperactivity disorder) diagnosed by a specialist physician in the field and according to Diagnosis and Statistics of Mental Disorders-5 (DSM-5) criteria.
* Subject of any psychotropic treatment for at least 15 days before inclusion
* Subject committing not to take any treatment during the study period, nor to participate in another therapeutic treatment in parallel.
* Subject available and pledging to honor the two weekly neurofeedback sessions for 15 consecutive weeks, and be available for symptom monitoring at 6 months.
* Child benefiting from a Social Security scheme.

Non Inclusion Criteria:

* Neurological disorders (epilepsy)
* Trouble of the autistic spectrum
* Active disorder without hyperactivity (TDA)
* Bad understanding of the French language
* Low Intellectual Level (IQ <70 Cognitive Assessment)
* Lack of understanding of the constraints inherent in the protocol
* Inability to comply with the constraints of the study throughout its duration

Exclusion Criteria:

* premature termination of participation, withdrawal of the patient's voluntary informed consent
* Investigator's or sponsor's decision
* Withdrawal of consent of subjects or legal guardians

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a neurofeedback protocol on the symptoms of Attention-Deficit with Hyperactivity Disorder (ADHD) | scores between baseline and after 15 weeks
  ADHD symptoms will be assessed using the clinician version of the 18-item Attention-Deficit with Hyperactivity rating scale IV (ADHD-RS). Each item is scored on a 0-3 scale with 0 representing the absence of the behavior/symptom and 3 representing the very frequent and impairing behavior/symptom over the last months. Two subscales compose ADHD-RS: 9-item Inattention subscale (range: 0-27) and a Hyperactivity-Impulsivity subscale (range: 0-27). The total ADHD-RS score is the sum of the two subscale scores and ranges from 0 to 54.
  Effectiveness of a neurofeedback protocol on the training capacity will be defined as a decrease of at least 30% the ADHD-RS total score between baseline, after 15 workout sessions of neurofeedback (2 sessions per week) and another 15 workout sessions of neurofeedback (2 sessions per week). Patients completing the study will therefore have undergone 30 workout sessions of neurofeedback

SECONDARY OUTCOMES:
Stability of change in ADHD symptoms after 6-month follow-up | scores between 15 weeks and after 6 months
  The ADHD-RS total score will be rated after a 6-month follow-up period of time to assess the stability of changes compared with the last workout session of neurofeedback. Stability is defined as absolute variation of 10% of the ADHD-RS total score.
Scores on Inattention and Hyperactivity-Impulsivity components of ADHD during a neurofeedback protocol | scores between baseline and after 7weeks and after 15 weeks
  The changes on the Inattention and Hyperactivity-Impulsivity subscores of the ADHD-RS will be described: baseline, after 15 workout sessions of neurofeedback (2 sessions per week) and after another 15 workout sessions of neurofeedback (2 sessions per week). We expect a significant diminution of either or both scores compared with baseline (repeated testing)..
Sleep quality during a neurofeedback protocol using a questionnaire | between baseline and after 15 weeks and after 6 months
  Sleep quality will be assessed by the 19-item Pittsburgh Sleep Quality Index (PSQI) questionnaire filled by the patient with support of his/her parents at baseline, after 15 workout sessions of neurofeedback, after another 15 workout sessions of neurofeedback and after a 6-month follow-up period of time. The first four items are open while the next 15 items are rated on a 0 to 3 scale. Seven component scores are generated and further added to provide an overall score ranging from 0 to 21, lower scores denoting a healthier sleep quality.
Executive functions rated during a neurofeedback protocol | scores between baseline and after 15 weeks and after 6 months
  Executive functions are assessed using the Behavioral Performance Evaluation Inventory questionnaire (BRIEF) at baseline, after another 15 workout sessions of neurofeedback and after a 6-month follow-up period of time. When possible, both the Parent and Teacher versions of the BRIEF are filled out.
  The BRIEF questionnaire counts 86 items groups in eight non-overlapping clinical scales (Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor) and two validity scales (Inconsistency and Negativity) and two validity scales. The clinical scales form two broader Indexes (Behavioral Regulation and Metacognition) and an overall score, the Global Executive Composite. Scale scores are converted to T-scores providing information about the child's individual scores relative to the scores of other respondents in the standardization sample
Clinical Improvement during a neurofeedback protocol and after 6-month follow-up | Evolution between baseline and after 15 weeks and after 6 months
  Clinical severity will be assessed at baseline using Guy's Global Clinical Impression scale (CGI-S).The clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Ratings range to 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
  Clinical improvement will be assessed at baseline, after 15 workout sessions of neurofeedback after 30 workout sessions of neurofeedback and after a 6-month follow-up period of time. The clinician rates how much the patient's illness has improved or worsened relative to a state at the beginning of the protocol. Ratings range to 1 (Very much improved) to 7 (Very much worse).
Computerized measures of attention and impulsivity during a neurofeedback protocol | at baseline, after 15 weeks and after 6months
  A task-oriented computerised assessment of attention-related problem, the Conners Continuous Performance Test 3rd Edition (CPT-3), will be performed at baseline, after 15 workout sessions of neurofeedback, after another 15 workout sessions of neurofeedback and after a 6-month follow-up period of time. Lasting 14 minutes of time, the CPT-3 provides objective information about inattentiveness, impulsivity, sustained attention, and vigilance. The patient's results are compared with a large normative sample of 1,400 subjects

CONTACTS AND LOCATIONS:
Overall Officials: Hervé MD CACI, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux pédiatriques de Nice CHU Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No